CLINICAL TRIAL: NCT00363688
Title: Treating Patients With a History of Non-Life Threatening Allergic Reaction to Penicillin With Penicillin: Is It Safe?
Brief Title: Treating Patients With a History of Non-Life Threatening Allergic Reaction to Penicillin With Penicillin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 756497
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 1997-12

CONDITIONS: Penicillin Allergy
Keywords: Non life threatening allergic reaction; oral challenge; penicillin; skin testing

INTERVENTIONS:
Drug: Penicillin test and challenge

SUMMARY:
The purpose of this study is to examine whether oral challenge with penicillin for patients with a known history of non-life threatening allergic reaction to penicillin is well-tolerated irrespective of skin-testing results

DETAILED DESCRIPTION:
Objective: To examine whether oral challenge with penicillin for patients with a known history of non-life threatening allergic reaction to penicillin is well-tolerated irrespective of skin-testing results long after the event occurred.

Methods: In this prospective, open-label, controlled, multi-clinical trial, 8702 individuals from primary care clinics were screened for penicillin allergy. 169 patients with a history of non-life threatening allergic reaction to penicillin, dating back at least 3 years, were recruited for study. Regardless of the response to penicillin skin testing, patients received the recommended daily dosage of penicillin and amoxicillin on two separate occasions. 2-6 years later a follow-up was conducted to assess the outcomes of further penicillin administration.

Results: 92.9% of the patients had an allergic reaction 6 years or longer before enrollment in the study. Of 272 challenges, 137 were skin-test positive with mild rash in 9 patients (6.6%), and 135 were skin-test negative with similar allergic reaction in 5 (3.7%) (P =.29). At follow-up, 3 of 55 patients (5.5%) who were given a full treatment course of penicillin developed mild skin eruption.

Conclusions: A positive penicillin skin testing of patients with a history of non-life threatening allergic reaction to penicillin occurring 3 years or longer from the event was not associated with a greater prevalence of adverse reactions to oral challenge with penicillin than a negative one. It is of importance to determine whether oral challenge can serve as a diagnostic procedure for this particular group of patients, thereby saving the need for prior penicillin skin testing.

ELIGIBILITY:
Inclusion Criteria:patients with a history of non-life threatening allergic reaction to penicillin, dating back at least 3 years -

Exclusion Criteria:Patients who had a life-threatening anaphylactic reaction to penicillin consisting of unconsciousness or anaphylaxis requiring life-resuscitation and those who had non-IgE mediated hypersensitivity reactions

-

Ages: 4 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-01; Study Completion 2004-05

PRIMARY OUTCOMES:
results of an oral challenge with penicillin (penicillin V) and amoxicillin

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Goldberg, MD, Principal Investigator — Allergy and Clinical Immunology Unit, Meir Medical Center, Kfar Saba, and Sackler Faculty of Medicine, Tel-Aviv University, Tel-Aviv, Israel
Locations (1):
- Meir Medical Center, Kfar Saba, Israel